CLINICAL TRIAL: NCT00421057
Title: The Effects of Combined Strength Training and Functional Endurance Exercise Regimen on Cancer-Related Fatigue and Physical Performance
Brief Title: Combined Strength Training and Functional Endurance Exercise Regimen on Cancer -Related Fatigue and Physical Performance
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0309
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer; Fatigue
Keywords: Breast Cancer; Cancer-Related Fatigue; Fatigue; Exercise; Strength Training; Endurance Exercise; Questionnaire; Survey
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Motor Activity | interventions — Surveys and Questionnaires; Karnofsky Performance Status

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Exercise Group: Taught to perform a specific regimen for strength-training and walking exercises.
  Interventions: Behavioral: Combined Strength Training and Functional Endurance Exercise
- Nonexercise Group: Follow usual routines of standard care but not taught to perform a specific regimen for strength-training and walking exercises; will keep record of any exercises done that are not a part of this study.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Combined Strength Training and Functional Endurance Exercise — Participants will be taught to stretch a Theraband as far as your arms or legs can stretch and the proper posture for walking for exercise. The Estimated Timed-Get-Up and Go test (ETGUPGo) and a 6-minute walk test will be performed to check your level of fatigue and physical ability.
  Groups: Exercise Group
Behavioral: Questionnaire — Questionnaires taking approximately 30 minutes total to complete.
  Other Names: Survey; Schwartz Fatigue Scale; Karnofsky Performance Scale; International Physical Activity Questionnaire; IPAQ
  Groups: Nonexercise Group

SUMMARY:
Primary Objective:

-Determine if a specific exercise regimen (combined strength training/functional endurance) reduces the level of fatigue among women with breast cancer while undergoing adjuvant or neoadjuvant chemotherapy treatment as compared to a control group.

Secondary Objectives:

* Determine if a specific exercise regimen (combined strength training/functional endurance) increases the overall ability to perform daily physical activities (ADLs) among women with breast cancer while undergoing adjuvant or neoadjuvant chemotherapy treatment as compared to a control group.
* Determine if a specific exercise regimen (combined strength training/ functional endurance) increases mobility in women with breast cancer while undergoing adjuvant or neoadjuvant chemotherapy treatment as compared to a control group.
* Determine if a specific exercise regimen (combined strength training/functional endurance) increases endurance in women with breast cancer while undergoing adjuvant or neoadjuvant chemotherapy as compared to a control group.

DETAILED DESCRIPTION:
Cancer-related fatigue has been described as the most common and troubling side effect of cancer and cancer treatment. Researchers want to see if a strength-training and walking exercise regimen may help reduce severe fatigue and increase patients' ability to perform activities of daily living.

If you agree to take part in this study, you will complete a questionnaire, provide contact information, and participate in 1 of 2 groups. For the questionnaire, you will be asked information about your age, ethnic origin, marital status, education, exercise habits, and cancer diagnosis. It should take about 5 minutes to complete. For the contact information, you will be asked to provide the name, address, and telephone number of someone to call in case of an emergency.

After completing the questionnaire and providing the contact information, you will be randomly assigned (as in the toss of a coin) to 1 of 2 groups. Participants in the exercise group will be taught to perform a specific regimen for strength-training and walking exercises. Participants in the nonexercise group will follow the usual routines of standard care but will not be taught to perform a specific regimen for strength-training and walking exercises. Participants in the nonexercise group will be asked to keep a record of any exercises that are done for the participant's personal regimen that are not a part of this study. You will have an equal chance of being assigned to either group.

All participants in this study will be asked to complete questionnaires (the Schwartz Fatigue Scale, Karnofsky Performance Scale, and the International Physical Activity Questionnaire [IPAQ]) in the Breast Center Clinic before beginning chemotherapy treatment. The Schwartz Fatigue Scale and IPAQ will also be completed after chemotherapy treatment. All of these questionnaires will be used to provide information about your physical activities and how much time you spend doing them. It should take about 25-30 minutes to complete all 3 questionnaires.

No matter what group you are in, after these questionnaires are completed, a physical therapist will then escort you to the exercise room located in the Physical Therapy and Rehabilitation Clinic. The therapist will perform a lymphedema (excess fluid collection) evaluation that will involve measuring the size of your arms and hands by placing a tape measure around your arms and hands at 5 different points. The lymphedema evaluation will be done at each clinic visit when you come in for chemotherapy and 2 weeks after completing your therapy. You will also be asked to complete exercise testing, the Estimated Timed-Get-Up and Go test (ETGUPGo) and a 6-minute walk test, to check your level of fatigue and physical ability. This exercise testing will be performed before you begin chemotherapy and within 2 weeks after you finish your last chemotherapy treatment. The exercise testing will be done after your chemotherapy treatment so that researchers can compare your level of fatigue and physical performance to what you were experiencing before your therapy began.

The ETGUPGo test will measure how fast you can rise from a chair, walk about 4 yards, turnaround and return to the chair, and sit down. For the 6-minute walk test the therapist will ask you to walk around in the exercise room at your own pace while the therapist counts the total time you were able to walk. Two (2) weeks after you have finished all of your treatments, you will re-take the Schwartz Fatigue Scale, Karnofsky Scale, IPAQ, ETGUPGo, and 6-minute walk test. Your exercise testing will be done in private, which means that no one other than the study staff will be allowed to enter the room while you are being tested.

If you are assigned to the group that will have a specific exercise regimen, you will be taught a strengthening and walking exercise. For the strengthening regimen, you will be taught to stretch a Theraband (material that looks like a big rubber band) as far as your arms or legs can stretch. You will be taught to perform this exercise at home. You will be able to look at pictures of these exercises in a booklet that will be provided to you. You will be asked to perform these exercises 3-5 times per week. For the walking regimen, you will be taught the proper posture for walking for exercise. You must walk at least once per day, but otherwise you may walk as often and as long as you feel like.

You will also have exercise testing. The therapist will measure the length of your arms and legs to see how much force it takes for you to stretch the rubber band beyond the length of your arms and legs. The therapist will test your current muscle strength by asking you to sit and rise from a chair, walk a certain distance, and return to the chair. You will also be asked to walk a certain distance until you get tired. The therapist will record how much time it takes you to complete both exercises (strengthening and walking).

After you begin the exercises at home, the research nurse will call you every 2 weeks and ask you how many times you performed the strengthening exercises throughout the week as well as the average amount of time you walked each day. The phone call should last about 10-15 minutes each time. You will be asked to check the box on an exercise calendar (that will be provided to you) showing which exercises you were able to perform each day.

All exercise testing will be given on the day of your routine visits to the clinic.

Your participation will be complete in this study after you perform your last exercise testing (about 2 weeks after your last chemotherapy treatment).

This is an investigational study. However, if you begin to experience some emotional distress that is directly related to this study, you may be referred for professional counseling here at M. D. Anderson in the Social Work Department. The social services staff will be available to assist you with the referral outside of the M. D. Anderson system. Up to 58 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a clinical diagnosis of breast cancer (Stages I - III),
2. be between the ages of 21 and 60 years;
3. may have undergone definitive surgical procedure (lumpectomy or mastectomy), and
4. be scheduled to receive any chemotherapy/hormonal blocker regimen that is appropriate for treatment of breast cancer (neoadjuvant or adjuvant)
5. approval of the Oncologist responsible for overseeing the cancer treatment plan for the patient to participate in this study.

Exclusion Criteria:

1. Exclusion criteria include presence of concomitant major health problems in which an exercise regimen is contraindicated (e.g. cardiac, pulmonary, and orthopedic)
2. Currently participating in a structured exercise program which is defined as a regular walking, stretching, and or dance type exercise that is performed at least 30 minutes or greater each time and more than 3 times per week.
3. Women who have had breast reconstructive surgery.
4. Men diagnosed with breast cancer.

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants with breast cancer that will be receiving chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Patient Fatigue Scores | Approximately 6 months
  Self-reported score that measures subjective perceptions of fatigue in which respondents rate their experience of feeling tired. It ranges from 1 (not at all) to 5 (extremely) and describes discomforts of cancer related fatigue in four dimensions (physical, mental, emotional, and temporal) (Schwartz and Meek, 1999).

CONTACTS AND LOCATIONS:
Overall Officials: Geneva Caldwell, MSN, RN, Principal Investigator — U.T. M.D. Anderson Cancer
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org